CLINICAL TRIAL: NCT05460130
Title: Implementation of a Simplified, Low-barrier Primary Care HCV Treatment Model for High Risk, High Prevalence Populations in Austin, Texas
Brief Title: Implementing HCV Treatment for High-risk Populations in Austin, Texas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Tim Mercer, Assistant Professor, Chief of the Division of Global Health, Departments of Population Health and Internal Medicine, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study 1656; IN-US-987-6016 (Other Grant/Funding Number: Gilead Sciences, Inc.)
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C Virus Infection
Keywords: DAAs; SVR12; Implementation Science; homelessness; direct-acting antivirals; sustained virological response; healthcare for the homeless; people who inject drugs
MeSH Terms: conditions — Hepatitis C | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Other): Persons infected with the hepatitis C virus who meet the study inclusion criteria and do not meet one or more of the exclusion criteria.
  Interventions: Behavioral: Simplified Hepatitis C Virus (HCV) Treatment Protocol

INTERVENTIONS:
Behavioral: Simplified Hepatitis C Virus (HCV) Treatment Protocol — A simplified, low-barrier, locally contextualized, HCV treatment protocol delivered by trained front-line health care providers (primary care physicians and mid-level providers) serving hard-to-reach-populations.

SUMMARY:
Highly-effective, pan-genotypic direct acting antivirals (DAAs) have made elimination of hepatitis C virus (HCV) a real possibility. A minority of the population infected with HCV has access to care or been prescribed such HCV treatment. Among people experiencing homelessness in the US, and seeking care at Health Care for the Homeless (HCH) clinics, prevalence is 31%, and 70% among people who experience homeless and inject drugs. In N. America, 55% of people who inject drugs (PWID) have HCV. Austin, TX has over 7,000 people experiencing homelessness with about 20% having a substance use disorder.

Treatment of HCV via DAAs is feasible and effective in primary care settings, and is as effective as treatment by specialists. Among people with opioid use disorder receiving opioid agonist therapy it's both effective and cost-effective. Treatment in the primary care setting has also been shown to be feasible and effective for people experiencing homelessness, with supporting evidence of engaging and retaining people in care. Furthermore, a novel HCV treatment model, featuring a simplified HCV treatment algorithm for front-line health care providers (primary care physicians, Nurse Practitioners, Physicians Assistants), has now been published, to help increase capacity, scale-up treatment and achieve elimination.

This study takes the foregoing new simplified approach one step further: Implementing this simplified algorithm for front-line health care providers in primary care settings caring for high-risk populations such as individuals experiencing homelessness and PWID. The novelty is providing treatment in diverse primary care settings, and targeting clinical sites serving high-risk populations, including people experiencing homelessness and PWID. Investigators use an implementation science approach to study the feasibility and effectiveness of the HCV treatment model in achieving HCV cure in high-risk populations.

Investigators hypothesize that by training front-line health care providers on a simplified, low-barrier HCV treatment model and adapting it using a locally contextualized, protocol-driven approach, investigators will effectively scale up HCV treatment across multiple primary care clinical sites serving high-risk populations, yielding sustained virologic response at 12 weeks (SVR-12) in 75% of enrolled participants. Investigators predict theHCV treatment model to measure favorably across implementation process and outcome measures of reach, adoption, implementation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18 years and older.
* Enrolled in care at one of CommunityCare's clinical sites participating in the study.
* Laboratory diagnosis of HCV
* Chronic hepatitis C infection

Exclusion Criteria:

* Have decompensated cirrhosis.
* Have received hepatitis C treatment previously.
* Had a liver transplant or actively on the transplant list awaiting a liver transplant.
* Have resistant HCV virus
* Infected with HIV
* Infected with hepatitis B
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with chronic HCV infection enrolled in the study that achieve SVR-12 | The measurement of SVR12 is assessed 12 weeks after completing treatment.
  A sustained virological response is defined as an undetectable HCV RNA level 12 weeks after treatment completion.

SECONDARY OUTCOMES:
Clinical outcome: Time to treatment | Approximately 10 months from time of enrollment
  Time elapsed (in days) from being offered treatment to initiating treatment
Clinical outcome: Complete HCV Treatment | Approximately 10 months from time of enrollment
  Proportion of participants enrolled in the study who complete HCV treatment
Clinical outcome: Initiate HCV treatment | Approximately 10 months from time of enrollment
  Proportion of participants enrolled in the study who initiate HCV treatment

OTHER OUTCOMES:
Implementation Outcome: Reach | Approximately one year from date of enrollment of first participant
  Proportion of participants with chronic HCV enrolled in the study who are offered treatment
Implementation Outcome: Adoption | Approximately one year from date of enrollment of first participant
  Proportion of clinical sites that adopt the HCV treatment protocol
Implementation Outcome: Implementation | Approximately one year from date of enrollment of first participant
  Qualitative interviews to assess the extent to which the HCV treatment protocol was implemented as intended (fidelity)
Implementation Outcome: Maintenance | Approximately one year from date of enrollment of first participant
  Qualitative interviews to assess the extent to which the HCV treatment protocol is sustained over time

CONTACTS AND LOCATIONS:
Overall Officials: Timothy I Mercer, MD,MPH, Principal Investigator — The University of Texas at Austin Dell Medical School; Darlene Bhavnani, PhD MPH, Principal Investigator — The University of Texas at Austin Dell Medical School
Locations (1):
- CommUnityCare Health Centers, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desai A, Reinis K, O'Neal L, Chang P, Brown C, Stefanowicz M, Kuang A, Agrawal D, Mercer T, Bhavnani D. Implementation of Site-Specific Hepatitis C Virus Treatment Workflows for Vulnerable, High-Risk Populations: A Prospective Single-Arm Trial. J Prim Care Community Health. 2025 Jan-Dec;16:21501319251330622. doi: 10.1177/21501319251330622. Epub 2025 Mar 31. PMID 40162901
- [Derived] Desai A, O'Neal L, Reinis K, Chang P, Brown C, Stefanowicz M, Kuang A, Agrawal D, Bhavnani D, Mercer T. Development, implementation, and feasibility of site-specific hepatitis C virus treatment workflows for treating vulnerable, high-risk populations: protocol of the Erase Hep C study - a prospective single-arm intervention trial. Pilot Feasibility Stud. 2023 May 8;9(1):78. doi: 10.1186/s40814-023-01311-4. PMID 37158965